CLINICAL TRIAL: NCT04916210
Title: Determinants of Incident Stroke Cognitive Outcomes and Vascular Effects on RecoverY
Acronym: DISCOVERY
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Natalia Rost, MD, Professor of Neurology, Massachusetts General Hospital
Other Study IDs: 2020P001099; U19NS115388 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-06-07 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Dementia, Vascular; Mild Cognitive Impairment; Vascular Cognitive Impairment
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Dementia, Vascular; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be collected from all participants at baseline for genomic and blood-based biomarker analyses. Tier 2 and 3 participants will undergo additional blood draws at each in-person follow-up visit for the collection of whole blood and RNA for longitudinal blood-based biomarker and DNA methylation (DNAm) analyses.
  Plasma, whole blood and RNA samples will be frozen and stored at the DISCOVERY Biorepository at the University of California, San Diego (UCSD) or the University of Southern California (USC) for further processing, storage and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of the DISCOVERY study is to better understand what factors contribute to changes in cognitive (i.e., thinking and memory) abilities in patients who experienced a stroke. The purpose of the study is to help doctors identify patients at risk for dementia (decline in memory, thinking and other mental abilities that significantly affects daily functioning) after their stroke so that future treatments may be developed to improve outcomes in stroke patients. For this study, a "stroke" is defined as either (1) an acute ischemic stroke (AIS, or blood clot in the brain), (2) an intracerebral hemorrhage (ICH, or bleeding in the brain), (3) or an aneurysmal subarachnoid hemorrhage (aSAH, or bleeding around the brain caused by an abnormal bulge in a blood vessel that bursts).

The investigators hypothesize that:

1. The size, type and location of the stroke play an important role in recovery of thinking and memory abilities after stroke, and pre-existing indicators of brain health further determine the extent of this recovery.
2. Specific stroke events occurring in individuals with underlying genetic or biological risk factors can cause further declines in brain heath, leading to changes in thinking and memory abilities after stroke.
3. Studying thinking and memory alongside brain imaging and blood samples in patients who have had a stroke allows for earlier identification of declining brain health and development of individualized treatment plans to improve patient outcomes in the future.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, nested-cohort study. A total of 8,000 patients hospitalized at the DISCOVERY clinical sites with acute-onset AIS, ICH or aSAH and no history of dementia will be enrolled.

All participants will undergo baseline screening for evidence of pre-stroke dementia. Those who pass baseline screening will complete a blood draw and a series of cognitive and functional assessments at baseline.

Participants will undergo in-person (3-6 months, 18 months) and telephone (annual) follow-up visits for the duration of the study to assess for longitudinal cognitive and functional outcomes. In addition to Tier 1 procedures, at each in-person follow-up visit, Tier 2 participants will also undergo brain MRI scanning, comprehensive cognitive assessment batteries and longitudinal blood collection; and Tier 3 participants will also complete a specialized imaging of the brain (amyloid- and tau-PET/CT scans), which is intended to identify special biomarkers of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Admitted to the enrolling clinical performance site (CPS) hospital with a diagnosis of acute ischemic stroke (AIS), intracerebral hemorrhage (ICH), or aneurysmal subarachnoid hemorrhage (aSAH)
3. Radiographic confirmatory evidence of: (1) AIS (based on a focal area of restricted diffusion on MRI), (2) non-traumatic primary ICH (based on evidence of acute parenchymal hemorrhage on CT or brain MRI) or (3) non-traumatic acute aSAH (based on evidence of subarachnoid hemorrhage on CT or MRI and evidence of aneurysm on CT angiography, MR angiography, or conventional catheter-based angiography)
4. Able to complete baseline visit in person or by phone within 6 weeks of stroke onset
5. Able to provide informed consent by self or proxy
6. Fluent in English or Spanish prior to stroke onset

Exclusion Criteria:

1. Documented history of pre-stroke dementia or fails dementia pre-screen
2. Concurrently enrolled into a study that is not approved under the DISCOVERY Co-Enrollment Policy
3. Unable to complete study protocol (advanced directives such as comfort measures only, or inability to complete the study due to severe medical/behavioral co-morbidities), as determined by physician investigator during screening process

   Additional exclusion criteria for Tier 2 participants:
4. Contraindication to MRI: presence of electrically, magnetically, or mechanically activated implants (such as cardiac pacemakers, cochlear implants, implanted pumps); or metallic clips in the brain

   Additional exclusion criteria for Tier 3 participants:
5. Age <50 years
6. Biologically female individuals who are pregnant or seeking to become pregnant
7. Known to have one of the following genetic conditions which can increase the risk of developing cancer: Cowden disease, Lynch syndrome, hypogammaglobulinemia, Wiskott-Aldrich syndrome, Down's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent (≤ 6 weeks) acute ischemic stroke, intracerebral hemorrhage or aneurysmal subarachnoid hemorrhage and no history of dementia.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in post-stroke cognitive impairment and dementia (PSCID) diagnosis status | Baseline to 48 months post-index stroke

SECONDARY OUTCOMES:
Change in cognitive function | Baseline to 3-6, 12, 18, 24, 36 and 48 months post-index stroke

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rost, MD, MPH, Principal Investigator — Massachusetts General Hospital; Steven Greenberg, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (31):
- United States (31):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - University of Colorado, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami Health System, Miami, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Health, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - UTHealth, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Contingent upon approval from the DISCOVERY Project Steering Committee and Sharing Subcommittee, or the NINDS (upon completion of the study), data, imaging and/or samples from consenting participants may be shared with other external researchers for future research. All identifiers and study-specific codes will be removed and assigned a second randomized identifier. The key linking each identifier to a study-specific code will be in the possession of the DISCOVERY Repository Core and will not be shared with external researchers.
  Upon completion of the study, the study database will be available to NINDS along with a data dictionary and all information needed to utilize the data in future research in accordance with the informed consent. De-identified genetic information derived from this study will be deposited in the US NIH genomic database (dbGAP and future iterations) and used for future research.

REFERENCES:
- See also: Official Website for the DISCOVERY Study — https://discoverystudy.org/